CLINICAL TRIAL: NCT01798212
Title: A Prospective Multi Center Case Controlled Trial on the Clinical Feasibility of a New Full Thickness Endoscopic Plication Device for Patients With GERD.
Brief Title: Prospective Trial on the Clinical Feasibility of a New Full Thickness Endoscopic Plication Device for Patients With GERD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PlicatorLinz
Record Dates: First submitted 2013-02-18; First posted 2013-02-25 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- full thickness gastroplication (Other)
  Interventions: Procedure: endoscopic full thickness plication

INTERVENTIONS:
Procedure: endoscopic full thickness plication
  Other Names: GERDx™

SUMMARY:
A prospective multi center case controlled trial on the clinical feasibility of a new full thickness endoscopic plication device for patients with GERD.

The primary objective of the present trial is to investigate, clinical feasibility of the GERDx™ device, evaluating surgical aspects, quality of life, and symptom sores. Secondary objective of the trail is to evaluate objective data before and after the procedure, using manometry and 24h impedeance measurement

ELIGIBILITY:
Inclusion Criteria:

Written informed consent; ≥ 18 years of age;

GERD documented by 24h ambulatory Multichannel Impedance-pH-Monitoring off antisecretory therapy and/or Gastroscopy by one or more of the following criteria:

* Total Number of Reflux Events ≥ 73/24h;
* DeMeester Score ≥ 14.7;
* Positive Symptom Index - SI ≥ 50% for Symptoms troublesome for the Patient with a Frequency of at least 3/24hrs; Macroendoscopically distinct mucosal breaks.

Exclusion Criteria:

Patients with known immunological dysfunction (advanced liver disease, HIV, hepatitis C virus infection), drug addiction;

≤ 18 years of age; Pregnancy and lactation; Previous extensive abdominal surgery; Previous esophageal or gastric surgery; Hiatal hernia >2cm; paraesophageal hernia; American Society of Anaesthesiologists physical status classification >II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life using the Gastrointestinal Quality of Life Index | change from baseline in Quality of Life at 3 months, one year and three years after the intervation

SECONDARY OUTCOMES:
lower esophageal sphincter pressure using oesophageal manometry | change from baseline in lower esophageal sphincter pressure at 3 months, one year and 3 years after the intervantion
DeMeester score, number of reflux events using 24h-ph-Impedancemeasurment | change from baseline in DeMeester score at 3 months, one year and 3 years after the intervantion

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Krankenhaus Barmherzige Schwestern, Linz
  - Krankenhaus Zell am See, Zell am See